CLINICAL TRIAL: NCT01594827
Title: Persistent MRSA Eradication Protocol (PMEP)
Brief Title: Persistent Methicillin Resistant Staphylococcus Aureus Eradication Protocol (PMEP)
Acronym: PMEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Case Western Reserve University (Other); Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00017536
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Cystic Fibrosis
Keywords: Methicillin-resistant Staphylococcus aureus; Vancomycin
MeSH Terms: conditions — Cystic Fibrosis | interventions — Rifampin; Trimethoprim; Sulfamethoxazole; Trimethoprim, Sulfamethoxazole Drug Combination; Doxycycline; Mupirocin; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled Vanc and Oral Abx (Experimental): In the experimental arm CF participants are randomized to 28 days of inhaled sterile vancomycin (250 mg twice a day) as well as 28 days of oral/skin antibiotics targeted to aggressively treat MRSA infection: oral rifampin, a second oral antibiotic (TMP/SMX or doxycycline, protocol determined), mupirocin intranasal cream and chlorhexidine body washes. Patients will be followed for 3 months after completion of the treatment protocol.
  Interventions: Drug: Inhaled Vancomycin; Drug: Rifampin; Drug: Trimethoprim/Sulfamethoxazole (TMP/SMX); Drug: Doxycycline; Drug: Mupirocin Intranasal Creme; Drug: 4% chlorhexidine gluconate liquid skin cleanser
- Inhaled Placebo and Oral Abx (Active Comparator): In the active comparator arm CF participants are randomized to 28 days of inhaled sterile placebo (saline) and are treated with 28 days of oral/skin antibiotics targeted to aggressively treat MRSA infection: oral rifampin, a second oral antibiotic (TMP/SMX or doxycycline, protocol determined), mupirocin intranasal cream and chlorhexidine body washes. Patients will be followed for 3 months after completion of the treatment protocol.
  Interventions: Drug: Placebo (Sterile Water); Drug: Rifampin; Drug: Trimethoprim/Sulfamethoxazole (TMP/SMX); Drug: Doxycycline; Drug: Mupirocin Intranasal Creme; Drug: 4% chlorhexidine gluconate liquid skin cleanser

INTERVENTIONS:
Drug: Inhaled Vancomycin — On Days 1-28, subjects will receive nebulized Vancomycin. This will be supplied as a 250 mg solution to be nebulized two times a day for 28 days in 5cc sterile water. Patients will use a Pari Sprint nebulizer and Pari Vios compressor as the delivery system.
  Other Names: Vanc
  Arms: Inhaled Vanc and Oral Abx
Drug: Placebo (Sterile Water) — On Days 1-28, subjects will receive 5cc of a nebulized Placebo (Sterile water) twice a day. This is a taste (quinine 0.1mg/mL) matched nebulized placebo (sterile water). Patients will use a Pari Sprint nebulizer and Pari Vios compressor as the delivery system.
  Other Names: Placebo
  Arms: Inhaled Placebo and Oral Abx
Drug: Rifampin — Oral Rifampin by mouth for 28 days
  1. >45 kg: 600 mg by mouth daily
  2. 35-45 kg : 450 mg by mouth daily
  3. 25-34.9 kg: 300 mg by mouth daily
  Other Names: Rifadin
Drug: Trimethoprim/Sulfamethoxazole (TMP/SMX) — Oral trimethoprim/sulfamethoxazole (DS-160/800)
  1. >45 kg: two DS tablets twice a day by mouth (320/1600)
  2. 25-45 kg: one DS tablet twice a day by mouth (160/800)
  Other Names: Bactrim; Septra
Drug: Doxycycline — If sulfa intolerant or TMP/SMX Resistant, use instead oral doxycycline
  1. >45 kg: 100 mg by mouth twice a day
  2. 35-45 kg : 75 mg by mouth twice a day iii. 25-34.9 kg: 50 mg by mouth twice a day
  Other Names: Vibramycin; Adoxa
Drug: Mupirocin Intranasal Creme — Mupirocin 2% intranasal creme: half of single use tube applied into each nostril twice a day for 5 days.
  Other Names: Bactroban
Drug: 4% chlorhexidine gluconate liquid skin cleanser — Hibiclens 15cc liquid skin cleanser packets (4% chlorhexidine gluconate): use three packets once weekly for four weeks in the shower from the neck to toes, with attention on the axilla, groin, and buttocks.
  Other Names: Hibiclens

SUMMARY:
The prevalence of methicillin resistant Staphylococcus aureus (MRSA) respiratory infection in Cystic Fibrosis (CF) has increased dramatically over the last decade. Evidence suggests that persistent infection with MRSA may result in an increased rate of decline in Forced Expiratory Volume (FEV)1 and shortened survival. Currently there are no conclusive studies demonstrating an effective aggressive treatment protocol for persistent MRSA respiratory infection in CF. Data demonstrating an effective and safe method of clearing persistent MRSA infection are needed.

The purpose of this study is to evaluate the safety and efficacy of a 28-day course of vancomycin for inhalation, 250 mg twice a day, (in combination with oral antibiotics) in eliminating MRSA from the respiratory tract of individuals with CF and persistent MRSA infection. Subjects will be assigned in a 1:1 ratio to either vancomycin for inhalation (250 mg twice a day) or taste matched placebo and will be followed for 3 additional months. In addition, both groups will receive oral rifampin, a second oral antibiotic (TMP-SMX or doxycycline, protocol determined), mupirocin intranasal cream and chlorhexidine body washes. Forty patients with persistent respiratory tract MRSA infection will be enrolled in this trial.

DETAILED DESCRIPTION:
Primary Objectives

The primary objectives of this trial are to:

1. Determine the efficacy of an aggressive treatment protocol in eradicating persistent MRSA infection in individuals with CF.
2. Determine the safety of an aggressive treatment protocol in eradicating persistent MRSA infection in individuals with CF.

Secondary Objectives

The secondary objectives of this trial are to:

1. Determine the efficacy of an aggressive treatment protocol in improving Forced Expiratory Volume (FEV)1, time to exacerbation, and quality of life in individuals with CF and persistent MRSA infection.
2. Determine if there is benefit to adding nebulized vancomycin to an aggressive oral antibiotic treatment protocol in eradicating persistent MRSA infection in individuals with CF.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 12 years of age.
2. Confirmed diagnosis of CF based on the following criteria:

   positive sweat chloride > 60 mEq/liter (by pilocarpine iontophoresis) and/or a genotype with two identifiable mutations consistent with CF or abnormal Nasal Potential Difference (NPD), and one or more clinical features consistent with the CF phenotype.
3. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.
4. Two positive MRSA respiratory cultures in the last two years at least six months apart, plus a positive MRSA respiratory culture at Screening Visit and Run-in (Day -14) Visit.
5. At least 50% of respiratory cultures from the time of the first MRSA culture (in the last two years) have been positive for MRSA.
6. Forced Expiratory Volume (FEV)1 > 40% of predicted normal for age, gender, and height at Screening, for subjects 18 years of age or older..
7. FEV1> 60% of predicted normal for age, gender, and height at Screening, for subjects 12--17 years of old.
8. Females of childbearing potential must agree to practice one highly effective method of birth control, including abstinence. Note: highly effective methods of birth control are those, alone or in combination, that result in a failure rate less than 1% per year when used consistently and correctly. Female patients who utilize hormonal contraceptives as a birth control method must have used the same method for at least 3 months before study dosing. If the patient is using a hormonal form of contraception, patients will be required to also use barrier contraceptives as rifampin can affect the reliability of hormone therapy. Barrier contraceptives such as male condom or diaphragm are acceptable if used in combination with spermicides

Exclusion Criteria:

1. An acute upper or lower respiratory infection, pulmonary exacerbation, or change in routine therapy (including antibiotics) for pulmonary disease within 42 days of the Day 1 Visit (2 weeks prior to Screening visit).
2. Individuals on chronic continuous inhaled antibiotics without interruption who are not willing to substitute vancomycin or placebo for their scheduled inhaled antibiotic during days 0-28 of the study (every other month inhaled antibiotics are acceptable)
3. Use of oral or inhaled anti-MRSA drugs within two weeks of the Screening Visit.
4. History of intolerance to inhaled vancomycin or inhaled albuterol.
5. History of intolerance to rifampin or both TMP/SMX and doxycycline.
6. Resistance to rifampin or both TMP/SMX and doxycycline at Screening.
7. Resistance to vancomycin at Screening.
8. Abnormal renal function, defined as creatinine clearance < 50 mL/min using the Cockcroft-Gault equation for adults or Schwartz equation in children, at Screening.
9. Abnormal liver function, defined as ≥ 3x upper limit of normal (ULN), of serum aspartate transaminase (AST) or serum alanine transaminase (ALT), or known cirrhosis. at the time of Screening.
10. Serum hematology or chemistry results which in the judgment of the investigator would interfere with completion of the study.
11. History of or listed for solid organ or hematological transplantation
12. History of sputum culture with non-tuberculous Mycobacteria in the last 6 months.
13. History of sputum culture with Burkholderia Cepacia in the last year.
14. Planned continuous use of soft contact lenses while taking rifampin and no access to glasses.
15. Current use of oral corticosteroids in doses exceeding the equivalent of 10 mg prednisone a day or 20 mg prednisone every other day
16. Administration of any investigational drug or device within 28 days of Screening or within 6 half-lives of the investigational drug (whichever is longer).
17. Patients on inhaled antibiotics must have been on the same regimen for the 4 months prior to screening
18. Female patients of childbearing potential who are pregnant or lactating, or plan on becoming pregnant
19. Any serious or active medical or psychiatric illness, which in the opinion of the investigator, would interfere with patient treatment, assessment, or adherence to the protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Boyle, MD, Principal Investigator — Johns Hopkins School of Medicine; James Chmiel, MD, Principal Investigator — Case Western University
Locations (2):
- United States (2):
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dasenbrook EC, Checkley W, Merlo CA, Konstan MW, Lechtzin N, Boyle MP. Association between respiratory tract methicillin-resistant Staphylococcus aureus and survival in cystic fibrosis. JAMA. 2010 Jun 16;303(23):2386-92. doi: 10.1001/jama.2010.791. PMID 20551409
- [Background] Dasenbrook EC, Merlo CA, Diener-West M, Lechtzin N, Boyle MP. Persistent methicillin-resistant Staphylococcus aureus and rate of FEV1 decline in cystic fibrosis. Am J Respir Crit Care Med. 2008 Oct 15;178(8):814-21. doi: 10.1164/rccm.200802-327OC. Epub 2008 Jul 31. PMID 18669817
- [Background] Jennings MT, Boyle MP, Weaver D, Callahan KA, Dasenbrook EC. Eradication strategy for persistent methicillin-resistant Staphylococcus aureus infection in individuals with cystic fibrosis--the PMEP trial: study protocol for a randomized controlled trial. Trials. 2014 Jun 12;15:223. doi: 10.1186/1745-6215-15-223. PMID 24925006
- [Derived] Lo DK, Muhlebach MS, Smyth AR. Interventions for the eradication of meticillin-resistant Staphylococcus aureus (MRSA) in people with cystic fibrosis. Cochrane Database Syst Rev. 2022 Dec 13;12(12):CD009650. doi: 10.1002/14651858.CD009650.pub5. PMID 36511181
- See also: Johns Hopkins Cystic Fibrosis Center website — http://www.hopkinscf.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Persistent MRSA Eradication Protocol (PMEP) was a double-blind, randomized, placebo-controlled study performed at two CF centers (Johns Hopkins Hospital, Baltimore, MD; and University Hospitals Rainbow Babies and Children's Hospital, Cleveland, Ohio.) The study was conducted from October 2012 through March 2017.
Pre-assignment Details: After qualifying for and enrolling in the study based on inclusion criteria, participants were required to again demonstrate MRSA positive respiratory culture at the run-in visit (day -14) in order to be randomized to treatment arms. 39 participants were assessed for eligibility but only 29 matched inclusion criteria and were randomized.
Groups:
- Inhaled Vancomycin and Oral Antibiotics: In the experimental arm CF participants were randomized to 28 days of inhaled sterile vancomycin (250 mg twice a day) as well as 28 days of oral/skin antibiotics targeted to aggressively treat MRSA infection: oral rifampin, a second oral antibiotic (TMP/SMX or doxycycline, protocol determined), mupirocin intranasal cream and chlorhexidine body washes. Patients were followed for 3 months after completion of the treatment protocol.
- Inhaled Placebo (Sterile Water) and Oral Antibiotics: In the active comparator arm CF participants were randomized to 28 days of inhaled sterile placebo (saline) and treated with 28 days of oral/skin antibiotics targeted to aggressively treat MRSA infection: oral rifampin, a second oral antibiotic (TMP/SMX or doxycycline, protocol determined), mupirocin intranasal cream and chlorhexidine body washes. Patients were followed for 3 months after completion of the treatment protocol.
Period: Overall Study
Arm/Group | Inhaled Vancomycin and Oral Antibiotics | Inhaled Placebo (Sterile Water) and Oral Antibiotics
Started | 14 | 15
Completed | 10 | 15
Not Completed | 4 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Inhaled Vancomycin and Oral Antibiotics: In the experimental arm CF participants are randomized to 28 days of inhaled sterile vancomycin (250 mg twice a day) as well as 28 days of oral/skin antibiotics targeted to aggressively treat MRSA infection: oral rifampin, a second oral antibiotic (TMP/SMX or doxycycline, protocol determined), mupirocin intranasal cream and chlorhexidine body washes. Patients will be followed for 3 months after completion of the treatment protocol.
- Inhaled Placebo (Sterile Water) and Oral Antibiotics: In the active comparator arm CF participants are randomized to 28 days of inhaled sterile placebo (saline) and are treated with 28 days of oral/skin antibiotics targeted to aggressively treat MRSA infection: oral rifampin, a second oral antibiotic (TMP/SMX or doxycycline, protocol determined), mupirocin intranasal cream and chlorhexidine body washes. Patients will be followed for 3 months after completion of the treatment protocol.
- Total: Total of all reporting groups
Arm/Group | Inhaled Vancomycin and Oral Antibiotics | Inhaled Placebo (Sterile Water) and Oral Antibiotics | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Median (Full Range); unit: years] | 25.5 [12 to 46] | 25.0 [14 to 38] | 25.0 [12 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 15 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29
MRSA positive at baseline [Count of Participants; unit: Participants] | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients MRSA Free by Induced Sputum Respiratory Tract Culture
Description: The hypothesis for our primary outcome is that the aggressive treatment arm will result in significantly greater eradication of persistent MRSA from the respiratory tract of CF adolescents and adults on day 58 (1 month after completion of therapy) compared to the placebo/standard treatment arm. Our primary outcome will be comparing the proportion of CF patients in the treatment arm who have a negative induced sputum MRSA culture at Day 58 to the proportion of patients in the placebo arm who have a negative induced sputum MRSA culture at Day 58.
Time Frame: Day 58 (Visit 5), approximately 1 month after completion of the MRSA treatment protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Vancomycin and Oral Antibiotics | Inhaled Placebo (Sterile Water) and Oral Antibiotics
Number analyzed (Participants) | 10 | 15
Participants | 2 | 3

2. Secondary Outcome: Percentage of Patients MRSA Free by Induced Sputum Respiratory Tract Culture
Description: Percentage of patients MRSA free by induced sputum respiratory tract culture one day after completion of four-week eradication protocol (Day 29) in intervention arm vs standard treatment arm
Time Frame: Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Vancomycin and Oral Antibiotics | Inhaled Placebo (Sterile Water) and Oral Antibiotics
Number analyzed (Participants) | 10 | 15
Participants | 5 | 6

3. Secondary Outcome: Change in Forced Expiratory Volume (FEV1)% Predicted From Baseline to Day 58
Description: Change in Forced Expiratory Volume (FEV1)% predicted from baseline to day number 58
Time Frame: Baseline, Day 58
Measure: Median (Inter-Quartile Range); unit: % predicted FEV1
Arm/Group | Inhaled Vancomycin and Oral Antibiotics | Inhaled Placebo (Sterile Water) and Oral Antibiotics
Number analyzed (Participants) | 10 | 15
% predicted FEV1 | -2.5 [-6.0 to 1.0] | 1.0 [-5.0 to 6.0]

4. Secondary Outcome: Time to First CF Exacerbation
Description: Time to First CF Exacerbation using a standardized exacerbation definition from Day 1 to Day 118
Time Frame: Day 1 to Day 118
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Inhaled Vancomycin and Oral Antibiotics | Inhaled Placebo (Sterile Water) and Oral Antibiotics
Number analyzed (Participants) | 10 | 15
Days | NA (NA) — No exacerbations occurred in this group | 68.4 (22.2)

5. Secondary Outcome: Total Number of Pulmonary Exacerbations
Description: Total Number of Pulmonary Exacerbations using a standardized exacerbation definition at Days 58 and Days 118 in treatment vs. standard care group
Time Frame: Days 58 and 118
Measure: Number; unit: Exacerbations
Arm/Group | Inhaled Vancomycin and Oral Antibiotics | Inhaled Placebo (Sterile Water) and Oral Antibiotics
Number analyzed (Participants) | 10 | 15
Exacerbations
  Day 58 | 0 | 1
  Day 118 | 0 | 3

6. Secondary Outcome: Change if FEV1% Predicted From Screening
Description: Change in FEV1% predicted from Screening at Days 29, 58, and 118 in treatment vs. standard care group
Time Frame: Days 29, 58, and 118
Measure: Mean (Standard Error); unit: FEV1% predicted
Arm/Group | Inhaled Vancomycin and Oral Antibiotics | Inhaled Placebo (Sterile Water) and Oral Antibiotics
Number analyzed (Participants) | 10 | 15
FEV1% predicted
  Day 29 | 0.0 (2.1) | 1.1 (2.5)
  Day 58 | -3.0 (2.1) | 1.3 (2.5)
  Day 118 | -2.1 (1.4) | -0.3 (2.2)

7. Secondary Outcome: Change in Patient Reported Quality of Life (CFQ-R)(Respiratory)
Description: Change in Patient Reported Quality of Life (CFQ-R)(respiratory) from baseline to Days 29 and 58. CFQ-R stands for Cystic Fibrosis Quality of Life Measure, Respiratory Domain. Overall range of absolute score 0 to +80. Higher score means better quality of life. Positive change in score means improvement in quality of life. Minimally clinically significant difference: +/- 4.0 units.
Time Frame: Days 29 and 58
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Inhaled Vancomycin and Oral Antibiotics | Inhaled Placebo (Sterile Water) and Oral Antibiotics
Number analyzed (Participants) | 10 | 15
units on a scale
  Day 29 | 3.3 (4.1) | 11.5 (4.2)
  Day 58 | -4.4 (5.0) | 3.2 (4.8)

8. Secondary Outcome: Development of Antibiotic Resistance
Description: Number of patients with newly developed MRSA resistance to vancomycin, TMP/SMX, doxycycline, or rifampin.
Time Frame: Day 58 (Visit 5)
Population: No resistance to doxycycline or TMP/SMX. All developed resistance was to rifampin.
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Vancomycin and Oral Antibiotics | Inhaled Placebo (Sterile Water) and Oral Antibiotics
Number analyzed (Participants) | 10 | 15
Participants | 3 | 3

9. Secondary Outcome: Time to First Anti-MRSA Antibiotics (After Treatment Period)
Description: Time between completion of Study Drug and need for anti-MRSA antibiotics to control or treat symptoms
Time Frame: Completion of Study Drug to Day 118
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Inhaled Vancomycin and Oral Antibiotics | Inhaled Placebo (Sterile Water) and Oral Antibiotics
Number analyzed (Participants) | 10 | 15
days | NA (NA) — There were no exacerbations requiring treatment in this group | 58 (15)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of enrollment until 3 months after completion of treatment.
Description: Adverse events were collected at each study visit as per protocol
Arm/Group | Inhaled Vancomycin and Oral Antibiotics | Inhaled Placebo (Sterile Water) and Oral Antibiotics
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/14 | 3/15
Other Adverse Events (participants affected / at risk) | 14/14 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Vancomycin and Oral Antibiotics (N=14) | Inhaled Placebo (Sterile Water) and Oral Antibiotics (N=15)
Pulmonary Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 3 — All events occurred in the follow-up period not while on active treatment
Bowel Obstruction (Gastrointestinal disorders) | 1 | 0 — Occurred in the follow-up period not while on active treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Vancomycin and Oral Antibiotics (N=14) | Inhaled Placebo (Sterile Water) and Oral Antibiotics (N=15)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Diarrhea (Gastrointestinal disorders) | 7 | 2
Throat Symptoms (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Chest Tightness (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Headache (Nervous system disorders) | 3 | 5
Nausea (Gastrointestinal disorders) | 4 | 2
Heartburn (Gastrointestinal disorders) | 2 | 4
Chest Pain (General disorders) | 3 | 2
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Drop in FEV1 (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Increase in Sputum Production (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Chest Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 3

LIMITATIONS AND CAVEATS:
Easy termination leading to smaller number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT01594827/Prot_SAP_000.pdf